CLINICAL TRIAL: NCT03084211
Title: A Randomized Controlled Trial Comparing Prescribed Light Exercise to Standard Management for Emergency Department Patients With Acute Mild Traumatic Brain Injury.
Brief Title: Prescribed Light Exercise for ED Patients With MTBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Principal Investigator, Catherine Varner, MD, Clinician Scientist, Mount Sinai Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MSHED002
Record Dates: First submitted 2017-03-13; First posted 2017-03-20 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Mild Traumatic Brain Injury
Keywords: emergency department; concussion; head injury
MeSH Terms: conditions — Brain Concussion; Emergencies; Craniocerebral Trauma

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The control group will be instructed to gradually return to activities.
- Prescribed Light Exercise Group (Experimental): Intervention: Prescribed Light Exercise Group will receive discharge instructions prescribing 30 minutes of light exercise (ie: walking).
  Interventions: Other: Light exercise discharge instructions

INTERVENTIONS:
Other: Light exercise discharge instructions — Participants in the intervention group will receive discharge instructions prescribing light exercise following mild traumatic brain injury.
  Arms: Prescribed Light Exercise Group

SUMMARY:
Introduction: Current guidelines for treating patients with mild traumatic brain injury (MTBI) recommend a period of cognitive rest and gradual return to usual activities with avoidance of any activity that exacerbates symptoms. However, recent studies have reported prolonged rest beyond 48 hours might hinder MTBI recovery, and there is limited evidence to suggest following guidelines has a positive impact on prognosis. Given the paucity of effective management strategies to prevent post-concussion syndrome (PCS) and emerging evidence of the benefits of exercise in MTBI patients, there is an urgent need for more research on the effectiveness of an early exercise intervention in the acute MTBI patient population as prevention of PCS.

Research Question: Among adult (18-64 years) patients presenting to the ED with a discharge diagnosis of acute MTBI (defined by the Zurich consensus statement), does prescribing light exercise (ie: 30 min daily walking) reduce the proportion of patients with PCS at 30 days, compared to standard discharge instructions?

Methods: This will be a randomized controlled trial of adult (18-64 years) patients discharged from an academic ED diagnosed with MTBI occurring within 48 hours of the index ED visit. The intervention group will receive discharge instructions prescribing 30 minutes of light exercise (ie: walking) and the control group will be instructed to gradually return to activities. Discharge instructions will be read by the attending physician or ED nurse. Patients will be provided a printed copy of the discharge instructions. Depending on their preferences, patients will be contacted by email or by telephone to complete the Rivermead Post-Concussion Symptoms Questionnaire (RPQ), a validated, 16 item questionnaire.

The primary outcome of this study will be the proportion of patients with PCS at 30 days, defined as an increase from baseline of ≥ 3 symptoms on the validated RPQ at 1 month. Secondary outcomes will include change in RPQ from baseline to 72 hours, 7 days, 14 days, 30 days post initial ED visit, number of missed days of school or work and repeat visits to a healthcare provider. To assess compliance with ED discharge instructions, patients will be asked to complete a daily activity journal and will be given fitness tracking devices.

DETAILED DESCRIPTION:
Introduction:The emergency department (ED) is the first point of health care contact for most head injured patients. The majority (estimated 85%) of patients suffering head injury will not have intra-cranial damage requiring neurosurgical consultation, but may have symptoms of mil traumatic brain injury (MTBI). Patients with MTBI may have physical, emotional, behavioral, or cognitive symptoms such as headache, sleep disturbance, disorders of balance, fatigue, irritability, memory and concentration problems, and the majority have self-limited symptoms that abate within 7 to 10 days. Although early and spontaneous resolution occurs in most patients, a small proportion of adults with MTBI will have a protracted course. It is estimated between 15-30% of patients with MTBI develop post-concussion syndrome (PCS), which is a persistence of head injury symptoms after MTBI.3 PCS usually lasts 2-4 months, and the symptoms typically peak 4-6 weeks following the injury4. However, in a smaller percentage of patients, the symptoms of PCS last for a year or longer. Approximately 20% of adults with PCS will not have returned to full-time work 1 year after the initial injury, and some are disabled permanently by PCS.

Current guidelines recommend a period of 'cognitive rest' and stepwise return to usual activities following MTBI. Cognitive rest is defined as the avoidance of mental activities that may trigger symptoms, such as watching television, using the computer, exercising, or talking on the phone. Patients following 'return to usual activity' instructions are encouraged to only resume normal activities once symptoms have resolved, and if symptoms return upon recommencement of activities, to return to rest. However, a recent systematic review of early educational interventions in the ED for MTBI concluded there are no clear and consistent interventions or standard management practices that exist for this population. Additionally, previous research evaluating a period of strict bed rest, which includes both physical and cognitive rest, has also not been shown to decrease severity or duration of MTBI symptoms. Based on the best available evidence, current guidelines for the management of MTBI suggest complete bed rest should be avoided after the first 48 hours post-injury.

Regular exercise has been shown to have positive effects on well-being, including mental health, improved self esteem, sleep and memory. Recent studies including patients with PCS have reported exercise treatment programs improved exercise tolerance and decreased symptoms, even for those patients where exercise previously exacerbated PCS symptoms. Additionally, Wise et al., randomized patients with severe TBI to either a structured exercise program for 10 weeks or usual care and found patients in the exercise group were less depressed and reported better health status compared to those not included in the exercise program.

Rationale: Given the paucity of effective management strategies that prevent PCS following MTBI and emerging evidence of the benefits of exercise in MTBI patients, there is an urgent need for more research on the effectiveness of an early exercise intervention in the acute MTBI patient population as prevention of PCS.

Research Question: Among adult (18-64 years) patients presenting to the ED with a discharge diagnosis of acute MTBI (defined by the Zurich consensus statement), does prescribing light exercise (ie: 30 min daily walking) reduce the proportion of patients with PCS at 30 days, compared to standard discharge instructions?

Methods:

Study Design and Population This randomized controlled trial will be conducted in the ED of an academic tertiary care hospital (annual census 60,000). Consecutive, adult (18-64 years) patients presenting to the ED with a MTBI sustained within the preceding 48 hours will be eligible for enrollment. Acute MTBI will be defined by the Zurich consensus statement as a direct blow to the head, face, neck or elsewhere on the body with a force transmitted to the head which may or may not involve loss of consciousness AND results in brain injury with 1 or more symptoms in 1 or more of the following clinical domains: somatic, cognitive, emotional or behavioral, or sleep.

Triage nurses will screen potential patients and once eligibility is confirmed by the attending physician, informed written consent will be obtained from trained research personnel (when available) or by the attending physician or nurse. The study protocol will be approved by the local institutional Research Ethics Board and registered with clinicaltrials.gov.

Trained research personnel will collect demographic and clinical parameters (history, physical examination findings, diagnostic testing, ED management) from paper and electronic charts using a standardized data collection tool. The research assistant will ask patients to complete an inventory of symptoms to establish a baseline using the Rivermead Post-Concussion Symptoms Questionnaire (RPQ), a validated, 16 item questionnaire and provide instructions to the patient regarding the wearable step counter.

Interventions After providing informed written consent, patients will be randomized to either discharge instructions prescribing 30 minutes of light exercise (ie: walking) daily (intervention) or discharge instructions describing graduated return to usual activities and cognitive rest (control) using a fixed 1:1 allocation ratio produced by a computer-based random number generator. Block sizes of four will be used to ensure equal allocation to each group. To avoid potential patient selection and allocation bias, all physicians, nurses, RAs and patients will be blinded to the randomization schedule.

Sealed, sequentially numbered, opaque envelopes will contain the pre-assigned group allocation. By necessity, the physician administering the instructions and the patient will be aware of their allocation. However, outcome assessors will be blinded to group assignment.

Prior to receiving the discharge instructions, all patients will complete the RPQ questionnaire. Patients will be contacted via telephone at 2, 4 and 6 weeks following their index ED visit to repeat the RPQ questionnaire and determine if they have any subsequent MTBI-related physician visits and how many days of work or school they have missed due to MTBI symptoms. If telephone contact is not successful on the first day of scheduled follow-up, participants will be sent a text message to remind them of the scheduled telephone interview. If contact is not made within this timeframe, patients will be considered lost to follow-up and their data will be excluded from further analysis.

Discharge instructions will be read by the attending physician or ED nurse. Patients will be provided a printed copy of the discharge instructions. All patients will receive instructions including a description of common symptoms following MTBI and warning signs for missed intracranial injury such as vomiting, stupor, focal weakness, seizure and severe headache. The control group discharge instructions have been adapted from the Centers for Disease Control and Prevention Acute Concussion Evaluation Care Plan (work version) for healthcare providers. These MTBI discharge instructions describe a graduated return to usual activities plan based on head injury symptoms and emphasized cognitive rest. The intervention group will receive discharge instructions prescribing 30 minutes of light exercise (ie: walking) and the control group will be instructed to gradually return to activities.

Outcome Measures The primary outcome of this study will be the proportion of patients with PCS at 30 days, defined as an increase from baseline of ≥ 3 symptoms on the validated RPQ at 1 month. Secondary outcomes will include change in RPQ from baseline to 72 hours, 7 days, 14 days, 30 days post initial ED visit, number of missed days of school or work and repeat visits to a healthcare provider. To assess compliance with ED discharge instructions, patients will be asked to complete a daily activity journal and will be given step counters.

Data Analyses Data will be entered directly into a study specific Microsoft Excel database (Microsoft Corporation, Redmond, Washington). Descriptive statistics will be summarized using means with standard deviations (SD), medians with interquartile ranges (IQR) or frequencies with 95% confidence intervals (CIs) where appropriate. Differences in RPQ at 72 hours, 7 days, 14 days, 30 days post ED visit between the intervention and control groups will be compared using paired samples t-tests. Other outcomes including included change in number of missed days of school or work, repeat visits to a healthcare provider, and quality of life indicators will be compared between groups using descriptive statistics with 95% confidence intervals where appropriate. Analyses will be conducted according to the intention-to-treat principle.

Additionally, the tracking devices' measurements will be compared to the patients' reported symptoms and reported daily activity. All statistical analyses will be conducted using SAS (v.9.4, SAS institute, Inc., Cary, NC, USA).

ELIGIBILITY:
Inclusion Criteria:

- MTBI occurring within 48 hours of the index emergency department visit

Exclusion Criteria:

* Acute intracranial injury identified on head CT
* Multisystem injuries prohibiting light exercise
* Existing medical condition that would compromise ability to participate in light exercise
* GCS < 15 at time of ED discharge
* Underlying neurological condition resulting in communication difficulties
* Insurmountable language barrier
* Inability to follow-up via telephone
* Alcohol or drug intoxication

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 367 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2019-10-03 (Actual); Study Completion 2019-10-03 (Actual)

PRIMARY OUTCOMES:
proportion of patients with PCS | 30 days
  Defined as an increase from baseline of ≥ 3 symptoms on the validated Rivermead Post-Concussion Symptoms Questionnaire

SECONDARY OUTCOMES:
Change in RPQ from baseline | 72 hours, 7 days, 14 days, 30 days post initial ED visit
  Between group differences of changes in RPQ will be compared.
Days of school or work missed | 72 hours, 7 days, 14 days, 30 days post initial ED visit
  Between group differences will be compared.
Return visits to a health care provider | 72 hours, 7 days, 14 days, 30 days post initial ED visit
  Between group differences will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Varner, MD MSc, Principal Investigator — Sinai Health System
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
No IDP will be shared with other researchers.

REFERENCES:
- [Derived] Varner CE, Thompson C, de Wit K, Borgundvaag B, Houston R, McLeod S. A randomized trial comparing prescribed light exercise to standard management for emergency department patients with acute mild traumatic brain injury. Acad Emerg Med. 2021 May;28(5):493-501. doi: 10.1111/acem.14215. Epub 2021 Feb 28. PMID 33481332